CLINICAL TRIAL: NCT05006456
Title: Real-world Experience of Catheter Ablation Using Novel Ablation Technologies Associated With the Carto System for the Treatment of Symptomatic Paroxysmal and Persistent Atrial Fibrillation (NOVEL AF)
Brief Title: Real-world Experience of Catheter Ablation Using Novel Ablation Technologies for the Treatment of Atrial Fibrillation
Acronym: NOVEL AF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Heart Health Research Center (Other); Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Chang sheng Ma, Prof., Beijing Anzhen Hospital
Other Study IDs: 2021-novel
Record Dates: First submitted 2021-07-14; First posted 2021-08-16 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Cohort 1 consists of 2000 subjects undergoing catheter ablation with STSF catheter, in which AI is used to guide the ablation lesion creation.
  Interventions: Device: Catheter ablation
- Cohort 2: Cohort 2 consists of 2000 subjects who undergoing catheter ablation using QDOT or HELIOSTAR catheter.
  Interventions: Device: Catheter ablation

INTERVENTIONS:
Device: Catheter ablation — Subjects will undergo catheter ablation using the new technologies, including THERMOCOOL SMARTTOUCH® SF catheter with Visitag SURPOINT, QDOT catheter and HELIOSTAR catheter when they are used in conjunction with Carto system for AF ablations.

SUMMARY:
The primary purpose of this registry is to obtain real-world clinical experience for the latest and future ablation technologies when used in conjunction with the Carto system in the treatment of patients with atrial fibrillation (AF) in Asian countries. The ablation technologies include THERMOCOOL SMARTTOUCH® SF (STSF) catheter with Ablation Index (AI) /Visitag SURPOINT, QDOT catheter, and HELIOSTAR catheter. Additional new ablation and/or mapping technologies may be included in future when they become available in local markets.

DETAILED DESCRIPTION:
Novel-AF study is a prospective, non-randomized, multi-center, longitudinal study.

1. Primary endpoint 1.1 The primary effectiveness endpoint is the percent of subjects who are freedom from atrial arrhythmia (any documented AF, atrial tachycardia (AT), or atrial flutter (AFL) episode of ≥30 seconds by heart rhythm monitoring patch, ECG, or Holter recording) from days 91 to 365 post ablation, with or without the use of any anti-arrhythmic drugs (AADs).

   1.2 The primary safety endpoint is the incidence of primary adverse events (PAEs), defined as procedure- or device-related serious adverse events occurred within 7 days of the procedure.
2. Secondary endpoint 2.1 Freedom from documented AF/AT/ AFL lasting≥30 seconds from days 91 to 365 post ablation without AADs 2.2 Acute procedural success of PVI, confirmed by entrance block in all pulmonary veins after adenosine and/or isoproterenol challenge 2.3 First pass isolation rate for STSF/QDOT and Single-Shot-Success (SSS) rate for HELIOSTAR per PV/ per patient before adenosine/isoproterenol challenge 2.4 Time to isolation (TTI) for HELIOSTAR per PV/ per patient before adenosine/isoproterenol challenge 2.5 Numbers of acute pulmonary vein (PV) reconnection after waiting/challenge, with number and location of any gaps in each patient 2.6 Procedural efficiency parameters [total procedure time, mapping time and points, LA time, fluoroscopy time and dose, RF application time per circle (left and right wide area circumferential ablation) and in total, needle time in transseptal puncture, and fluid volume delivered via catheter]
3. Follow up Follow-up visits will be scheduled at 3, 6, 9 and 12 months after the index ablation procedure 3.1 Subject baseline information: age, sex, height, weight, medical and heart surgery history, left ventricular ejection fraction (LVEF), left atrial dimension, left atrium volume, New York Heart Association (NYHA) Class, physical activity (IPAQ-S-CBaecke et al), depression (PHQ-9) and anxiety (PHQ-GAD-7), AF symptoms/duration, quality of life (AFEQT/EQ-5D), concomitant medications, LAA detection methods (CT/TEE/ICE), and results of laboratory tests 3.2 Peri-procedural data :

   * Procedural and ablation data: total procedure time, LA time, fluoroscopy time and dose, RF application time per circle
   * Ablation strategies: Ablation sites and the AI values for each ablation line
   * Acute success data
   * VISITAG® source database
   * Postprocedural complications/adverse events: device- and/or procedure-related serious adverse events (SAEs]
   * Periprocedural medications: anticoagulants, AADs, and sedation medicine
   * Duration of hospital stay. 3.3 Follow-up data
   * Patient information（details）
   * Concomitant medications
   * Any documented AF recurrence in 12-lead ECG, Holter, or any qualified monitoring equipment.
   * Re-ablation and ablation sites (if applicable)
   * Emergency room visit or hospitalization due to arrhythmia recurrence or procedure-related complications
   * New onset medical conditions
   * Adverse events

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Signed informed consent to participate in the study
* Drug refractory symptomatic paroxysmal AF or symptomatic persistent AF for less than 12 months who, in the opinion of the investigator, are candidates for catheter ablation per standard-of-care
* Undergoing AF ablation for the first time
* THERMOCOOL SMARTTOUCH® SF catheter with Visitag SURPOINT or newer technologies (e.g. QDOT, HELIOSTAR) are used in conjunction with Carto system in the ablation procedure

Exclusion Criteria:

* Women of childbearing potential who are, or plan to become, pregnant during the time of the study
* The subject has a life expectancy of less than 12 months
* Severe valvular heart disease
* The subject has been enrolled in another investigational study evaluating a medical device or a drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of adults age 18 years or older with symptomatic Paroxysmal and Persistent Atrial Fibrillation who are candidates for ablation
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
The percent of subjects who are freedom from atrial arrhythmia (any documented AF, atrial tachycardia (AT), or atrial flutter (AFL) episode. | 12 months
  percent of subjects who are freedom from atrial arrhythmia (any documented AF, atrial tachycardia (AT), or atrial flutter (AFL) episode of ≥30 seconds by heart rhythm monitoring patch, ECG, or Holter recording) from days 91 to 365 post ablation, with or without the use of any anti-arrhythmic drugs (AADs).
Incidence of primary adverse events (PAEs) | 7 days
  PAEs defined as procedure- or device-related serious adverse events occurred within 7 days of the procedure

SECONDARY OUTCOMES:
AF recurrence | 12 month
  Freedom from documented AF/AT/ AFL lasting≥30 seconds recording post ablation from days 91 to 365 without AADs, monitoring with ECG; Holter; Heart Rhythm Monitoring Patch;Dual/ CRT Pacer or ICD.
Acute procedural success of PVI | During ablation procedure
  Acute procedural success of PVI, confirmed by entrance block in all pulmonary veins after adenosine and/or isoproterenol challenge
First pass isolation rate | During ablation procedure
  First pass isolation rate for STSF/QDOT before adenosine/isoproterenol challenge
Single-Shot-Success (SSS) rate | During ablation procedure
  Single-Shot-Success (SSS) rate for HELIOSTAR per PV/ per patient before adenosine/isoproterenol challenge
Time to isolation (TTI) | During ablation procedure
  Time to isolation (TTI) for HELIOSTAR per PV/ per patient before adenosine/isoproterenol challenge
Proportion of acute pulmonary vein (PV) reconnection | During ablation procedure
  Proportion of acute pulmonary vein (PV) reconnection, with number and location of any gaps in each patient
Procedure time | During ablation procedure
  Including total procedure time，LA time，RF application time per circle ，needle time in transseptal puncture
Mapping points | During ablation procedure
  mapping points
fluid volume | During ablation procedure
  fluid volume delivered via catheter